CLINICAL TRIAL: NCT01285388
Title: A Dose Double-blind,Placebo-controlled,Single Dosing,Dose-escalation Clinical Trial to Investigate the Safety,Tolerability and Pharmacokinetic Characteristics of MB12066 in Healthy Male Subjects
Brief Title: Safety, Tolerability and Pharmacokinetic Study of MB12066 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yungjin Pharm. Co., Ltd. (Industry)
Collaborators: KT&G Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: MB12066_001
Record Dates: First submitted 2010-07-04; First posted 2011-01-28 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: Safety; Tolerability; Pharmacokinetic
MeSH Terms: conditions — Metabolic Syndrome; Obesity | interventions — beta-lapachone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- MB12066 10mg (Experimental)
  Interventions: Drug: MB12066
- MB12066 30mg (Active Comparator)
  Interventions: Drug: MB12066
- MB12066 100mg (Active Comparator)
  Interventions: Drug: MB12066
- MB12066 150mg (Active Comparator)
  Interventions: Drug: MB12066
- MB12066 200mg (Active Comparator)
  Interventions: Drug: MB12066
- placebo (Placebo Comparator)
  Interventions: Drug: MB12066

INTERVENTIONS:
Drug: MB12066 — MB12066 10mg, 100mg/tab. once oral dose MB12066 10, 30, 100, 150, 200mg
  Other Names: beta-lapachone

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of MB12066 after a single oral dose and to investigate the pharmacokinetic characteristics of MB12066 after a single oral dose.

DETAILED DESCRIPTION:
* Safety/ Tolerability evaluation

  -Adverse events, Physical examinations, Vital signs, ECG (including continuous ECG monitoring), Laboratory tests (including hematology, chemistry, coagulation, PBS, NAD(P)+/NAD(P)H ratio, urinalysis), CIC
* Pharmacokinetic Evaluation

  * Serial blood samples and urine collections for pharmacokinetic evaluations will be conducted between 0 (pre-dose) and 96 hours after a single oral dose.
  * Blood sampling time pre-dose, 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 36h, 48h, 72h post-dose
  * Urine collection time 0h - 6h, 6h - 12h, 12h - 24h, 24h - 48h, 48h - 72h
  * Evaluation parameters AUClast, AUCinf, Cmax, Tmax, t1/2, Vd/F, CL/F, Ae, fe, CLR

ELIGIBILITY:
Inclusion Criteria:

1. Subject is informed of the investigational nature of this study and voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB) - approved informed consent prior to performing any of the screening procedures
2. Healthy Korean male volunteers, age ranged 20 to 45 years (both inclusive)
3. A subject with body weight between 60 kg (inclusive) and 90 kg (exclusive) and body mass index (BMI) between 18.5 (inclusive) and 25 (exclusive). ☞ BMI (kg/m2) = weight (kg) / {height (m)}2
4. Findings within the range of clinical acceptability in medical history and physical examination, and laboratory results within the laboratory reference ranges for the relevant laboratory tests (unless the investigator considers the deviation to be irrelevant for the purpose of the study)

Exclusion Criteria:

1. A subject with history of allergies including drug allergies (aspirin, antibiotics, etc.), or history of clinically significant allergies
2. A subject with clinical evidence or history of hepatic (including carrier of hepatitis virus), renal, respiratory, endocrine, neurologic, immunologic, hematologic, oncologic, psychiatric, or cardiovascular disease
3. A subject with history of gastrointestinal disease or surgery (except simple appendectomy or repair of hernia), which can influence the absorption of the study drug
4. A subject whose hemoglobin(Hb) level < 12 g/dL
5. A subject with fasting plasma glucose (FPG) level ≤ 70 mg/dL or ≥ 126 mg/dL
6. A subject with HbA1c level ≥ 7.0 mmol/L
7. A subject whose systolic blood pressure (SBP) ≤ 90 mmHg or ≥ 140 mmHg, diastolic blood pressure (DBP) ≤ 40 mmHg or ≥ 90 mmHg or pulse rate (PR) ≥ 100 /min after at least 5 min sitting
8. A subject with history of drug abuse or positive urine drug screening test
9. A subject who has taken any prescribed medication or herbal compounds within 14 days prior to the study drug administration. In addition, a subject who has taken any over-the-counter drug or vitamin supplements within 7 days prior to the study drug administration (However, investigators can judge the subject, who has taken the medications during those periods above, eligible for the trial if all other conditions are satisfied.)
10. A subject who has participated in any other clinical trial either for investigational or marketed drugs within 8 weeks before the study drug administration
11. A subject who has donated or had loss of ≥ 400 mL of blood within 8 weeks prior to start of administration of study drug
12. A subject who consumes more than 21 units of alcohol per week or unable to stop drinking throughout the study period.
13. A smoker (except for whom quitted smoking prior to the drug administration for at least 3 months)
14. A subject who heavily takes caffeine or caffeine-containing products, grapefruit, grapefruit juice, grapefruit-containing products
15. A subject with unusual dietary habit
16. A subject who was previously assigned to treatment during this study
17. The investigator judges the subject not eligible for the study after reviewing clinical laboratory results or other reasons.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety/ Tolerability evaluation | from day-1 to day8-10
  Adverse events, Physical examinations, Vital signs, ECG (including continuous ECG monitoring), Laboratory tests (including hematology, chemistry, coagulation, PBS, NAD(P)+/NAD(P)H ratio, urinalysis), CIC

SECONDARY OUTCOMES:
Pharmacokinetic Evaluation | between 0 (pre-dose) and 96 hours after a single oral dose.
  * Blood sampling time pre-dose, 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 36h, 48h, 72h post-dose
  * Urine collection time 0h - 6h, 6h - 12h, 12h - 24h, 24h - 48h, 48h - 72h
  * Evaluation parameters AUClast, AUCinf, Cmax, Tmax, t1/2, Vd/F, CL/F, Ae, fe, CLR

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, Professor, Principal Investigator — Clinical Research Institute of Seoul National University Hospital